CLINICAL TRIAL: NCT04824677
Title: Risk Factors and Prognoses in Patients Hospitalized for COVID-19
Status: Completed | Type: Observational
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Ferran Barbe, Chair Respiratory Medicine, Sociedad Española de Neumología y Cirugía Torácica
Other Study IDs: COVID-Ponent
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — 1 tube EDTA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hospital treatment of COVID disease — Hospital treatment of COVID disease

SUMMARY:
Multicenter and observational study. The study will include patients admitted to hospitals in the Lleida health region with confirmed COVID-19. Follow-up will be carried out up to six months after hospital discharge.

Through the analysis of clinical data and biological parameters, it is possible to identify in advance patients who will evolve in an unfavorable prognosis in relation to COVID-19, either because they present criteria of severe disease or because they present thrombotic complications associated with the disease. The final aim is to make anticipated and individualized therapeutic decisions that reduce the morbidity and mortality associated with the disease.

DETAILED DESCRIPTION:
The main objective is to develop a predictive model of adverse events in hospitalized COVID-19 patients (death, initiation of mechanical ventilation, ICU admission and thrombotic event). An additional analyses will be performed for each individualized outcome.

Metodology: Prospective case-only study. The variables that will be collected are:

1. Previous epidemiological data of the patient.
2. Clinical and biological data and treatment upon admission to the hospital.
3. Clinical and biological evolutionary data (Increases in the values of certain biological variables in a defined period of time (> 48 h) during admission):

   * Baseline epidemiological and clinical variables
   * Baseline biological variables
   * Complications and clinical evolutionary variables
   * Evolutionary biological variables
4. Clinical evolutionary data of final outcomes, including death (at 30, 90 days and at 6 months), initiation of mechanical ventilation, ICU admission and thrombotic event.
5. For future studies of new biological and epigenetic variables, blood samples will be collected from hospitalized patients under the CIBER coverage.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed COVID-19 infection.
* Hospitalization in a center in the Lleida healthcare region.

Exclusion Criteria:

* Patients admitted with repeatedly negative COVID-19 test results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the participating centers of the Lleida health region, with a positive laboratory diagnosis for COVID19.
Sampling Method: Probability Sample
Enrollment: 971 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Composite endpoint (death, initiation of mechanical ventilation, ICU admission and thrombotic event) | 18 months
  Development of a predictive model of adverse events (death, initiation of mechanical ventilation, ICU admission and thrombotic event).

SECONDARY OUTCOMES:
Death | 18 months
  Development of a predictive model for mortality risk.
Mechanical ventilation | 18 months
  Development of a predictive model for the need of mechanical ventilation.
ICU admission | 18 months
  Development of a predictive model for admission at the ICU.
Thrombotic event | 18 months
  Development of a predictive model for the risk of thrombotic events.

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbé, MD, Principal Investigator — Spanish Respiratory Society (SEPAR)
Locations (2):
- Spain (2):
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitari Santa Maria, Lleida

REFERENCES:
- [Derived] Belmonte T, Perez-Pons M, Benitez ID, Molinero M, Garcia-Hidalgo MC, Rodriguez-Munoz C, Gort-Paniello C, Moncusi-Moix A, Made A, Devaux Y, Martelli F, Ortega A, Gonzalez J, Torres G, Barbe F, de Gonzalo-Calvo D. Addressing the unsolved challenges in microRNA-based biomarker development: Suitable endogenous reference microRNAs for SARS-CoV-2 infection severity. Int J Biol Macromol. 2024 Jun;269(Pt 2):131926. doi: 10.1016/j.ijbiomac.2024.131926. Epub 2024 Apr 28. PMID 38688344